CLINICAL TRIAL: NCT05250674
Title: Clinical Evaluation of CEM-guided Biopsy
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-8890
Record Dates: First submitted 2021-12-02; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2021-11

CONDITIONS: Contrast Enhanced Mammography-guided Biopsy
Keywords: Contrast Enhanced Mammography; breast cancer; interventional breast procedures
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Adult women with indication for a breast biopsy procedure after an abnormal CEM or MRI examination.: Adult women presenting with clinical indication for a breast biopsy procedure after a positive abnormal CEM or MRI examination and no clear ultrasound or mammography correlation.
  Interventions: Device: CEM-guided biopsy

INTERVENTIONS:
Device: CEM-guided biopsy — The evaluation population consists of adult women, presenting with clinical indication for a breast biopsy procedure after a positive abnormal CEM or MRI examination (with no clear ultrasound or mammography correlation) and considered eligible for this procedure as per standard of care.
  Eligible subjects undergo the clinically indicated breast biopsy procedure using the Pristina Serena Bright ® CEM-guided biopsy. Region of interest location is determined by using stereotactic pairs of CEM images after injection of iodinated contrast media. All necessary equipment and instrumentation, medications, or other devices required to complete the subject's clinically indicated procedure shall be used and are not expected to be influenced by evaluation participation.

SUMMARY:
CEM-guided biopsy is an optional accessory of Senographe Pristina intended to provide accurate location of lesions in the breast in three dimensions, using information obtained from Contrast Enhanced Mammography (CEM) images. This information provides guidance for a variety of minimally invasive or interventional procedures in the breast such as vacuum assisted biopsy, core biopsy, presurgical localization (e.g. hook wire), and fine needle aspirations (FNA). This device cannot be used for reasons other than its intended use.

This evaluation is being done to learn more about the CEM-guided biopsy. Clinical user and operational feedback is a central part of the development process for medical devices in which information from real clinical use is required to optimize the device prior to commercial release.

DETAILED DESCRIPTION:
Pristina Serena CEM is an option to the standard Pristina Serena breast biopsy unit. It is designed to allow the accurate localization of lesions in the breast in three dimensions, using information obtained from Contrast Enhanced Mammography (CEM) images. It is intended to provide guidance for histological purposes such as core or vacuum-assisted biopsies, for pre-surgical localization procedures, or Fine Needle Aspiration (FNA) for cytopathology analysis.

The main purpose of this evaluation is to collect feedback to assess image readability and look-and feel, usability, workflow and user preference information from physicians and technologists who use CEM-guided biopsy to perform minimally invasive interventional breast procedures under clinical conditions. All feedbacks are collected by observations, interviews and surveys.

The evaluation population consists of adult women, presenting with clinical indication for a breast biopsy procedure after a positive abnormal CEM or MRI examination, and considered eligible for this procedure as per standard of care.

Eligible subjects undergo the clinically indicated breast biopsy procedure using the Pristina Serena CEM-guided biopsy. Region of interest location is determined by using stereotactic pairs of CEM images after injection of iodinated contrast media. All necessary equipment and instrumentation, medications, or other devices required to complete the subject's clinically indicated procedure shall be used and are not expected to be influenced by evaluation participation.

ELIGIBILITY:
Inclusion Criteria:

* Adult women presenting with clinical indication for a breast biopsy procedure after a positive abnormal CEM or MRI examination, and considered eligible for this procedure as per standard of care.
* Are able and willing to comply with study procedures
* Are able and willing to provide written informed consent to participate

Exclusion Criteria:

* Findings not accessible for stereotactic guidance biopsy
* Are currently lactating
* Have breast implants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult women presenting with clinical indication for a breast biopsy procedure after a positive abnormal CEM or MRI examination, and considered eligible for this procedure as per standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Image visibility of enhancing finding | immediately after each CEM-guided biopsy
  To assess the visibility of an index enhancing finding at the point of the CEM-guided biopsy. The enhancement in the biopsy images will be compared to the enhancing lesion initially detected at the diagnostic CEM examination, that led to the prescription of the breast biopsy. It is a subjective and dichotomous measure: visible or not visible.

SECONDARY OUTCOMES:
Pathology results on biopsy specimen | up to 3 weeks
  Pathology results are classified according to the National Health Service Breast Screening Program (NHSBSP) classification for breast biopsies in B1 (normal tissue), B2 (benign lesion), B3 (lesion of uncertain malignant potential), B4 (suspicious), B5 (malignant).
Upgrade rate to malignancy of biopsied lesions that underwent surgical or percutaneous intervention | an average of 3 months
  To evaluate the upgrade rate to malignancy of lesions that were further assessed with surgical or percutaneous intervention. The term "upgrade to malignancy" applies for lesions that were diagnosed as high-risk lesions at biopsy (B3), but with final pathology at excision changed to malignancy (in situ or invasive), as well as for in situ lesions at biopsy upstaged to invasive cancer at surgery.
Number of participants with CEM-guided biopsy minor complications. | immediately after each CEM-guided biopsy
  To register the number of participants that underwent minor complications related to the CEM-guided procedure, such as presence of immediate hematoma in biopsy bed or experienced vasovagal reactions during or inmediately after the procedure. This information will be registered in three categories: hematoma, vasovagal reaction or no complications.
Biopsy needle approach | immediately after each CEM-guided biopsy
  To register the needle entry to the breast in order to access the intended lesion during the biopsy procedure as it was through a vertical or horizontal approach. It is a dichotomous measure: vertical or horizontal.
Total time per procedure | immediately after each CEM-guided biopsy
  To register the time spent during the biopsy procedure. The time will be considered since the intravenous contrast administration until the breast decompression, immediately after clip marker deployment. It is a numeric variable and will be measured in minutes and evaluated as a median interquartile range.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar - Parc de Salut Mar, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schrading S, Distelmaier M, Dirrichs T, Detering S, Brolund L, Strobel K, Kuhl CK. Digital breast tomosynthesis-guided vacuum-assisted breast biopsy: initial experiences and comparison with prone stereotactic vacuum-assisted biopsy. Radiology. 2015 Mar;274(3):654-62. doi: 10.1148/radiol.14141397. Epub 2014 Nov 11. PMID 25386875
- [Background] Wecsler J, Jeong YJ, Raghavendra AS, Mack WJ, Tripathy D, Yamashita MW, Sheth PA, Hovanessian Larsen L, Russell CA, MacDonald H, Sener SF, Lang JE. Factors associated with MRI detection of occult lesions in newly diagnosed breast cancers. J Surg Oncol. 2020 Mar;121(4):589-598. doi: 10.1002/jso.25855. Epub 2020 Jan 26. PMID 31984517
- [Background] Meissnitzer M, Dershaw DD, Lee CH, Morris EA. Targeted ultrasound of the breast in women with abnormal MRI findings for whom biopsy has been recommended. AJR Am J Roentgenol. 2009 Oct;193(4):1025-9. doi: 10.2214/AJR.09.2480. PMID 19770325
- [Background] Abe H, Schmidt RA, Shah RN, Shimauchi A, Kulkarni K, Sennett CA, Newstead GM. MR-directed ("Second-Look") ultrasound examination for breast lesions detected initially on MRI: MR and sonographic findings. AJR Am J Roentgenol. 2010 Feb;194(2):370-7. doi: 10.2214/AJR.09.2707. PMID 20093598
- [Background] Perlet C, Heywang-Kobrunner SH, Heinig A, Sittek H, Casselman J, Anderson I, Taourel P. Magnetic resonance-guided, vacuum-assisted breast biopsy: results from a European multicenter study of 538 lesions. Cancer. 2006 Mar 1;106(5):982-90. doi: 10.1002/cncr.21720. PMID 16456807
- [Background] Siegmann-Luz KC, Bahrs SD, Preibsch H, Hattermann V, Claussen CD. Management of breast lesions detectable only on MRI. Rofo. 2014 Jan;186(1):30-6. doi: 10.1055/s-0033-1335972. Epub 2013 Jul 29. PMID 23897532
- [Background] Santiago L, Candelaria RP, Huang ML. MR Imaging-Guided Breast Interventions: Indications, Key Principles, and Imaging-Pathology Correlation. Magn Reson Imaging Clin N Am. 2018 May;26(2):235-246. doi: 10.1016/j.mric.2017.12.002. Epub 2018 Feb 21. PMID 29622128
- [Background] Esserman LE, Cura MA, DaCosta D. Recognizing pitfalls in early and late migration of clip markers after imaging-guided directional vacuum-assisted biopsy. Radiographics. 2004 Jan-Feb;24(1):147-56. doi: 10.1148/rg.241035052. PMID 14730043
- [Background] Clauser P, Mann R, Athanasiou A, Prosch H, Pinker K, Dietzel M, Helbich TH, Fuchsjager M, Camps-Herrero J, Sardanelli F, Forrai G, Baltzer PAT. A survey by the European Society of Breast Imaging on the utilisation of breast MRI in clinical practice. Eur Radiol. 2018 May;28(5):1909-1918. doi: 10.1007/s00330-017-5121-4. Epub 2017 Nov 22. PMID 29168005
- [Background] Schrading S, Strobel K, Keulers A, Dirrichs T, Kuhl CK. Safety and Efficacy of Magnetic Resonance-Guided Vacuum-Assisted Large-Volume Breast Biopsy (MR-Guided VALB). Invest Radiol. 2017 Mar;52(3):186-193. doi: 10.1097/RLI.0000000000000331. PMID 27861232
- [Background] Neeter LMFH, Raat HPJF, Alcantara R, Robbe Q, Smidt ML, Wildberger JE, Lobbes MBI. Contrast-enhanced mammography: what the radiologist needs to know. BJR Open. 2021 Nov 24;3(1):20210034. doi: 10.1259/bjro.20210034. eCollection 2021. PMID 34877457